CLINICAL TRIAL: NCT03008707
Title: Laparoscopic Peritoneal Lavage vs Laparoscopic Sigmoidectomy in Perforated Acute Diverticulitis: a Multicenter Prospective Observational Study
Brief Title: Laparoscopic Peritoneal Lavage vs Laparoscopic Sigmoidectomy in Perforated Acute Diverticulitis: a Multicenter Prospective Observational Study (STELLA Study)
Acronym: STELLA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Ospedale San Jacopo, Pistoia (Unknown); S. Andrea Hospital (Other); Maggiore Bellaria Hospital, Bologna (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Hospitales Universitarios Virgen del Rocío (Other); George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Dario Tartaglia, MD, PhD Candidate, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: n° 890
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Acute Diverticulitis
Keywords: Laparoscopic peritoneal lavage; laparoscopic sigmoidectomy; complicated acute diverticulitis; D004238

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1: Patients who undergo Laparoscopic Peritoneal Lavage
  Interventions: Procedure: Laparoscopic Peritoneal Lavage
- Group 2: Patients who have a laparoscopically approached sigmoidectomy

INTERVENTIONS:
Procedure: Laparoscopic Peritoneal Lavage — LPL is done by irrigation with at least 6 L of warm saline throughout the abdominal cavity and after that, putting a drain in Douglas cavity through the port sites
  Groups: Group 1

SUMMARY:
Laparoscopic peritoneal lavage (LPL) has recently been emerging as an effective alternative to laparoscopic sigmoidectomy (LS) in patients with complicated acute diverticulitis (CAD) (Modified Hinchey's classification grade II non-responder to conservative therapy and grade III). Aim of the study is to evaluate which surgical strategy, between LPL and LS, could give better results in patients with CAD

DETAILED DESCRIPTION:
In the literature, there is no consensus about the role of the laparoscopic peritoneal lavage in the management of complicated acute diverticulitis. Recently, three important prospective randomized-control studies (SCANDIV, LOLA, DILALA) have reported contradicting conclusions, as two of them (SCANDIV and LOLA) state that LPL is not superior to sigmoidectomy for the high reoperation rate and morbidity, while DILALA confirms that LPL is feasible and safe in the short-term. To our knowledge, no international guidelines promote the use of LPL in complicated acute diverticulitis. We believe this technique could be safely used in a selected cohort of patients and, in some circumstances, could represent a "bridge" to a possible planned resection. The aim of the study is to collect and analyze the multicentric data of the LPL and LS and give a substantial contribution to the scientific community about this very debated topic.

ELIGIBILITY:
Inclusion Criteria:

* Acute abdominal pain,
* Signs of localized or diffuse peritonitis
* Signs of suspected perforated diverticulitis (diagnostic imaging)
* Signed informed consent

Exclusion Criteria:

* Septic shock
* Immunodepression
* Previous multiple abdominal surgical operations
* Modified Hinchey's grade IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complicated acute diverticulitis
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dario Tartaglia, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero, Universitaria Pisana, Pisa, Tuscany, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Laparoscopic Peritoneal Lavage: Patients who undergo Laparoscopic Peritoneal Lavage
  Laparoscopic Peritoneal Lavage: LPL is done by irrigation with at least 6 L of warm saline throughout the abdominal cavity and after that, putting a drain in Douglas cavity through the port sites
- Laparoscopically Approached Sigmoidectomy: Patients who have a laparoscopically approached sigmoidectomy
Period: Overall Study
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Started | 28 | 38
Completed | 28 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy | Total
Number analyzed (Participants) | 28 | 38 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.25 (13.21) | 55.68 (10.81) | 57.19 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 13 | 26 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 38 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Short-term Morbidity
Time Frame: 30 days
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 8 | 1

2. Primary Outcome: Short-term Mortality
Time Frame: 30 days
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 0 | 0

3. Primary Outcome: Optimal Sepsis Control
Time Frame: 30 days
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 19 | 37

4. Primary Outcome: Post-operative Re-interventions Rate
Time Frame: 15 days
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 5 | 0

5. Secondary Outcome: Mean Postoperative Time
Time Frame: 1 day
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
minutes | 76.74 (33.18) | 225.36 (81.58)

6. Secondary Outcome: Average Length of Postoperative Hospital Stay
Time Frame: 30 day
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
days | 11.4 (9.60) | 8.23 (5.21)

7. Secondary Outcome: Recurrent Colonic Diverticulitis Rate
Time Frame: 6 months
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 6 | 0

8. Secondary Outcome: Incisional Hernia Rate
Time Frame: 6 months
Population: In Laparoscopic Peritoneal Lavage, 1 patient out of 28 was excluded because of conversion to open surgery and resection
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
Number analyzed (Participants) | 27 | 38
Participants | 2 | 9

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Laparoscopic Peritoneal Lavage | Laparoscopically Approached Sigmoidectomy
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/38
Other Adverse Events (participants affected / at risk) | 0/27 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03008707/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03008707/SAP_001.pdf